CLINICAL TRIAL: NCT04315753
Title: Circulating and Imaging Biomarkers to Improve Lung Cancer Management and Early Detection
Acronym: SMAC-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Ospedale San Raffaele (Other); University of Paris 5 - Rene Descartes (Other); European Institute of Oncology (Other); Istituto Superiore di Sanità (Other)
Responsible Party: Sponsor
Other Study IDs: 1874
Record Dates: First submitted 2019-01-10; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer
Keywords: Biomarkers; Circulating tumor cells; Screening; Computer Tomography (CT Scan)
MeSH Terms: conditions — Lung Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cancer patients (clinical stage I and II) +controls: 70 lung cancer patients (clinical stage I and II) diagnosed outside screening and candidates to surgical resection at Humanitas Hospital, and 70 controls with benign nodules. Cancer patients will undergo blood collection before and at 4 months after surgical resection. Blood will be used for CTC analysis, exosome antigens and circulating free DNA (cfDNA) mutational analysis.
- prospective screening cohort of high risk individuals: a prospective screening cohort of high risk individuals enrolled at Humanitas Hospital (1000) will allow to recruit 50 patients with screening detected lung cancer and a large number of negative controls. Analysis of CTC, exosome antigens and cfDNA mutation profile will be performed.
  Interventions: Other: LDCT (Low Dose CT)

INTERVENTIONS:
Other: LDCT (Low Dose CT) — validate the role of non-invasive molecular and cellular biomarkers and combined radiomic signature, as complementary tools to assist early detection of lung cancer by LDCT using bioinformatic techniques for the integration of the results
  Other Names: Molecular biomarkers; Cellular biomarkers
  Groups: prospective screening cohort of high risk individuals

SUMMARY:
Validation of biomolecular markers in the circulation and radiomic features are the focus of this project.The aim is to assess the role of molecular and cellular biomarkers (exosomes antigens, Circulating tumor cells - CTCs, panel of mutations in circulating free DNA) and radiomic signature, as complementary to assist early detection of lung cancer by LDCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years old and exposure to smoking more than 30 packs-year; which corresponds to 6-year risk of lung cancer, calculated according to the plco score (≥ 2%).
* Smoker or former smoker Former smokers must have ceased smoking within the 15 years prior to enrollment in the study.
* Absence of symptoms of lung cancer such as worsening of cough, hoarseness, hemoptysis and weight loss.

Exclusion Criteria:

* Previous diagnosis of lung cancer.
* Positive extrapulmonary cancer history in the last 5 years (excluding in situ tumors or skin epidermoid tumor).
* Performing a chest CT scan in the last 18 months.
* Severe lung or extrapulmonary diseases that may preclude or invalidate appropriate therapy in case of diagnosis of malignant pulmonary neoplasia.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population should have the following inclusion criteria: Inclusion Criteria: - Age ≥ 55 years old and exposure to smoking more than 30 packsyear; which corresponds to 6-year risk of lung cancer, calculated according to the plco score (≥ 2%). - Smoker or former smoker Former smokers must have ceased smoking within the 15 years prior to enrollment in the study. - Absence of symptoms of lung cancer such as worsening of cough, hoarseness, hemoptysis and weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Obtaining biological samples, and correspondent clinical and imaging data to use, as fresh blood tissues or frozen stored tissues from lung cancer patients and controls obtained from the Division of Thoracic Surgery and LDCT lung-cancer screening program | 01 Jan 2018 - 01 Jan 2023
  1.1 : Obtaining biological material from cancer cases and controls (clinical cases) and store in the biobank with clinical data and imaging for bio radiomic analysis.
  1.2 : Identification and testing of methods of recruiting high-risk individuals for a lung-cancer screening program using available database to select very high risk individuals; 1.3 : Obtaining biological material from asymptomatic screening-detected cancer cases and controls and store in the biobank with clinical data and imaging.
  1.4 : Assessment of compliance of the recruited population and assessment of mean lung-cancer risk. Verify the potential impact of molecular markers as a pre-screening test to better assess the risk of subjects, evaluate the impact on nodule management and number of false positive cases among screening process according to biostatistical analysis.

SECONDARY OUTCOMES:
Tumor antigens identified by RPPA in lung cancer circulating exosome | 01 Jan 2018 - 01 Jan 2023
  Blood-derived exosomes will be collected. Exosome antigens assessment will be performed. Then, a bioinformatics analysis of the performance of exosome antigens as diagnostic markers for lung cancer will be performed.
Investigate the potential role of CTCs as diagnostic and prognostic tool in a screening content | 01 Jan 2018 - 01 Jan 2023
  3.1 Samples collection and preparation: isolation and count of CTCs; 3.2 Evaluation of diagnostic role of CTCs in early stage lung cancers; 3.3 Evaluation of the prognostic value of the number of CTCs at diagnosis (measured in terms of "progression free survival" and "overall survival"); 3.4 Characterization of CTCs for the expression of EMT and correlation with angiogenesis pattern of primary tumor; 3.5 Biostatistical analysis of the results.
Development and validation of a panel of mutations on circulating DNA as diagnostic test for lung cancer. | 01 Jan 2018 - 01 Jan 2023
  4.1 Samples collection and library preparation; 4.2 Standardisation of the technique; 4.3 Assessment of diagnostic role of the protein signature; 4.4 Bioinformatics analysis of the performance of the cell free DNA mutation signature as diagnostic tool for lung cancer
Investigate a radiomic signature to discriminate malignant lung nodule Background | 01 Jan 2018 - 01 Jan 2023
  5.1 assess the association of imaging features with clinical data and histology; 5.2 Identification the radiomic signature, the combination of imaging features, able to characterize lung lesions; 5.3 Validation of the signature on a new subset of patients; 5.4 Assessment of the role of radiomic signature, together with circulating markers in predicting lung malignancy

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No